CLINICAL TRIAL: NCT00224172
Title: Ambulatory Care Characteristics as Predictors of Mortality and Re-Admission
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Mary E. Charlson, MD, Weill Cornell Medical College
Other Study IDs: 0306006224 (Formerly 0603-908)
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2008-03-28 (Estimated); Status verified 2008-03

CONDITIONS: Ambulatory Care Patients Who Were Hospitalized in 2001 at the Cornell Campus of the New York-Presbyterian Hospital
Keywords: Pre-hospitalization characteristics; Post-hospitalization characteristics; Psychosocial measures; Predict re-hospitalization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to construct a prognostic model to identify risks of poor outcomes at one year following hospital discharge of patients treated in an ambulatory cate setting. The study will incorporate pre-hospitalization characteristics, hospitalization events, comorbidity burden, psychosocial measures and post-hospitalization care characteristics to predict re-hospitalization and mortality at one year.

DETAILED DESCRIPTION:
This model will identify potentially modifiable variables in the post-hospitalization clinic setting that result in increased rates of hospital readmission and mortality. Specifically, it is hypothesized that longer time to first outpatient visit after hospitalization, multiple providers, poor follow-up with scheduled appointment and discrepancies between discharge and outpatient medication lists will be predictors of adverse outcomes. Utilizing statistical modeling methods, it will be possible to recognize at risk patients, to identify modifiable risk factors and outpatient care characteristics, and in the future, to direct patient specific interventions to improve outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. All patients admitted to New York Presbyterian Hospital and followed in Cornell Internal Medicine Associated for at least one year prior to admission.

Exclusion Criteria:

1. Patients who do not wish to participate in the study.
2. Patients who are not followed in Cornell Internal Medicine Associates.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302
Dates: Start 2001-01; Study Completion 2001-12

PRIMARY OUTCOMES:
Psychosocial measures

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Charlson, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- New York Presbyterian Hospital-Weill Cornell Medical College, New York, New York, United States